CLINICAL TRIAL: NCT05896943
Title: The Application of Transcriptomics for Establishing Potential Prognostic Markers of Response to Treatment of Ulcerative Colitis With Ustekinumab
Brief Title: The Application of Transcriptomics in the Treatment of Ulcerative Colitis With Ustekinumab
Status: Completed | Type: Observational
Sponsor: Evangelismos Hospital (Other)
Responsible Party: Principal Investigator, Nikos Viazis, Consultant Gastroenterologist, Chief Department of Gastroenterology, Evangelismos General Hospital of Athens, Athens, Greece, Evangelismos Hospital
Other Study IDs: 479/15-12-2022
Record Dates: First submitted 2023-05-08; First posted 2023-06-09 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Ustekinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ulcerative colitis patients treated with ustekinumab: Patients with Ulcerative Colitis treated with ustekinumab
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — Patients with ulcerative colitis treated with ustekinumab

SUMMARY:
The investigators hope that the present study will highlight new transcriptomic prognostic markers of response to Ustekinumab with the ultimate goal of individualizing treatment and making a more targeted selection of UC patients who will benefit from this biological agent.

DETAILED DESCRIPTION:
Introduction: Optimizing treatment with biological agents is an ideal goal for patients with ulcerative colitis (UC). At present, there are insufficient prognostic markers of response to each biological agent, which makes it difficult to individualize treatment. Recent data suggest that mucosal inflammation patterns and serum cytokine profiles differ between patients who respond and those who do not. These studies mainly focused on anti-TNFα agents and Vedolizumab, while there are no corresponding data for Ustekinumab, which is a monoclonal antibody to interleukins 12 and 23 and has recently been approved for the treatment of patients with UC.

Aim of the study: To highlight prognostic markers of response (clinical and endoscopic) to Ustekinumab, in patients with UC, utilizing information from their transcriptome before starting treatment.

Methods: This is a prospective, single-center cohort study that will evaluate transcriptomic markers of response to Ustekinumab in patients with active UC. The diagnosis of the disease will be based on the established clinical, endoscopic and histological criteria. The patients' recruitment will begin in April 2022, while their consent will be required. The duration of follow-up of patients will be at least 6 months from the start of biological treatment. Patients will undergo endoscopy (sigmoidoscopy or total colonoscopy) with a biopsy of the orthosigmoid before the start of biological treatment and a repeat endoscopy 6 months later. The RNA profile of the patients will be recorded after isolation of the total RNA from colon biopsies. Then, using biostatistics, the transcriptomic profiles of patients who responded to Ustekinumab and those who did not respond to 6 months of treatment, will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Active UC in accordance with applicable diagnostic criteria [25] •
* Aged 18 or above

Exclusion Criteria:

* Prior surgical history for UC
* Toxic megacolon
* Infectious complications (Cl. Difficile, CMV infection)
* Patients who received any approved biologic agent (e.g. Infliximab, adalimumab, vedolizumab, golimumab) within the previous 8 weeks or any investigational biologic or other agent in the last 35 days

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Ulcerative Colitis treated with Ustekinumab
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
the rate of clinical remission | 6 months
  Total Mayo score of 2 or lower and no subscore higher than 1

SECONDARY OUTCOMES:
Endoscopic response rate | 6 months
  Reduction of the endoscopic Mayo subscore ≥1
Clinical response rate | 6 months
  Reduction in the Mayo score of at least 3 points and a decrease of at least 30% from the baseline score, with a decrease of at least 1 point on the rectal bleeding subscale or an Absolute rectal bleeding score of 0 or 1
Endoscopic remission rate | 6 months
  Endoscopic Mayo subscore 0

CONTACTS AND LOCATIONS:
Locations (1):
- Evangelismos Hospital, Athens, Attica, Greece